CLINICAL TRIAL: NCT01006434
Title: Weight Approximation in Stroke Before Thrombolysis
Acronym: WAIST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Martin Köhrmann, MD, University of Erlangen-Nürnberg Medical School
Other Study IDs: DE-ER-WAIST
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Stroke
Keywords: Stroke; Thrombolysis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Thrombolysis group (Pilot phase): Patients receiving intravenous thrombolysis for acute ischemic stroke. Pilot phase (100 Patients).
  Interventions: Other: Recording of body weight estimations, approximations and tPA dose
- Thrombolysis group: Patients receiving intravenous thrombolysis for acute ischemic stroke.
  Interventions: Other: Recording of body weight estimations, approximations and tPA dose

INTERVENTIONS:
Other: Recording of body weight estimations, approximations and tPA dose — Body weight estimation, patients are weighed, actual tPA dose is recorded

SUMMARY:
Thrombolysis using Alteplase (tPA) is still the only approved specific therapy for acute ischemic stroke (AIS). Current guidelines in western countries recommend an tPA dose of 0.9mg/kg up to a maximum dose of 90mg for patients weighing more than 100kg. However, larger dose-finding rtPA trials for intravenous thrombolysis in AIS are missing. Based on results from research on myocardial infarction only a few open label studies with low case rates were initiated to evaluate the optimal dose for tPA in cerebral ischemia. These studies suggested a narrow therapeutic range with decreased efficacy in lower dosages and an increased risk for thrombolysis related intracerebral hemorrhage (ICH) at doses above 0.95mg/kg. The ECASS-1 trial which used a dosage of 1.1mg/kg rt-PA showed significantly higher rate of large parenchymal hemorrhages compared to trials using 0.9mg/kg. Therefore accurate dosing is crucial. In the acute phase two aspects complicate rtPA dosing in AIS: First, unlike in other diseases many stroke patients are unable to communicate information on their body weight (BW) because of their stroke symptoms (e.g. aphasia, decreased consciousness). In addition motor symptoms prohibit easy weighing procedures in many patients. Second, the ultra-early and narrow time window for treatment does not allow time loss to weigh each patient in the emergency situation. Therefore routinely the attending physician has to make a visual estimation of the patient's BW. This may be inaccurate and may cause dosing errors which has been shown for other weight based emergency medication. There is little data on tPA-dosing errors in stroke patients and prospective data are lacking. The aim of our study is to evaluate availability of BW-information, accuracy of estimations and final dosing of tPA in a routine clinical setting. Therefore the investigators evaluate different sources of body weight estimations and also compare visual estimation with recently proposed anthropometric measurements for body weight approximation. Finally, impact of dosing errors on safety and efficacy are analyzed.

The initial phase will consist of 100 enrolled patients as a pilot phase for further power calculations. Based on the results of the pilot phase enrollment will continue. The envisioned inclusion target is up to 800 patients.

ELIGIBILITY:
Inclusion Criteria:

* all patients receiving intravenous thrombolysis with tPA for acute ischemic stroke

Exclusion Criteria:

* common exclusion criteria for intravenous thrombolysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving intravenous thrombolysis for acute ischemic stroke.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2008-04; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Dose dependent efficacy of thrombolysis. Modified Rankin Score after 3 Months. | 90 days
Dose dependent safety of thrombolysis | 90 days

SECONDARY OUTCOMES:
Availability and accuracy of body weight information. | 24 h
Accuracy of body weight estimations (medical personnel, patients) | 24 h
Dosage errors of tPA | 24 h

CONTACTS AND LOCATIONS:
Overall Officials: Martin Köhrmann, MD, Principal Investigator — Universityhospital Erlangen; Dept. of Neurology
Locations (1):
- Universityhospital Erlangen, Dept. of Neurology, Erlangen, Bavaria, Germany

REFERENCES:
- [Derived] Breuer L, Nowe T, Huttner HB, Blinzler C, Kollmar R, Schellinger PD, Schwab S, Kohrmann M. Weight approximation in stroke before thrombolysis: the WAIST-Study: a prospective observational "dose-finding" study. Stroke. 2010 Dec;41(12):2867-71. doi: 10.1161/STROKEAHA.110.578062. Epub 2010 Nov 11. PMID 21071723